CLINICAL TRIAL: NCT06592716
Title: Specificity and Sensitivity of Circulating HPV-DNA in Patients With Oropharyngeal Squamous Cell Carcinoma
Brief Title: Can Recurrence of Cancer in the Oropharynx be Detected by Blood Samples?
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Christian Grønhøj Larsen, Senior Registrar, PhD, DMSci, Assistant Professor, Rigshospitalet, Denmark
Other Study IDs: H-23071576; p-2023-15163 (Other: Capital Region of Denmark)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Oropharynx Cancer; Oropharynx Cancer, Metastatic; Oropharynx Cancer, Recurrent; Oropharyngeal Carcinoma; Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Keywords: HPV; HPV-DNA; Liquid biopsy; cell-free HPV-DNA; circulating HPV-DNA; circulating tumor HPV-DNA; ctHPV-DNA
MeSH Terms: conditions — Oropharyngeal Neoplasms; Neoplasm Metastasis; Recurrence; Squamous Cell Carcinoma of Head and Neck | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Liquid biopsies, in form of blood samples from peripheral veins
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Identify recurrence: The aim is to identify recurrence through longitudial analyses of circulating tumor HPV-DNA (ctHPV-DNA ) from blood samples.
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — The intervention is a liquid biopsy as a blood sample taken in a peripheral vein. The blood samples are analyzed for ctHPV-DNA.

SUMMARY:
This study investigates if longitudinal analyses of cell-free HPV-DNA in blood samples can be utilized to detect recurrence in patients diagnosed and treated for HPV-positive oropharyngeal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed HPV+ (and/or p16+) oropharyngeal squamous cell carcinoma
* Above 18 years of age
* Informed consent

Exclusion Criteria:

* The patient does not speak or understand Danish
* patients recieving palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HPV+ (and/or p16+) oropharyngeal squamous cell carcinoma
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of HPV ddPCR | At enrollment and at 2 months after end treatment, and hereafter every 6 month for a minimum of 2 years, up to 3 years, or at suspicion of recurrence.
  Sensitivity and specificity of the ddPCR ctHPV-DNA test compared to clinically or radiologically verified recurrence.

SECONDARY OUTCOMES:
Time to recurrence by ctHPV-DNA | From enrollment and for minimum 2 years, up to 3 years, after treatment
  Time to recurrence detected by ctHPV-DNA
Time to recurrence by clinical/radiological examination | From enrollment and for minimum 2 years, up to 3 years, after treatment
  Time to recurrence detected by clinical or radiological examination
PET/CT | From enrollment and for minimum 2 years, up to 3 years, after treatment
  Number of PET/CT scans without detectable recurrence
Cancer fast-track referrals | From enrollment and for minimum 2 years, up to 3 years, after treatment
  Number of referrals to Cancer Fast-track clinical investigations (conducted by an ENT specialist) without any detectable recurrences.
Fear of Recurrence Questionnaire | at 2 months after treatment, and hereafter every 6 months for a minimum of 2 years, up to 3 years
  Quality of Life (QoL) will be evaluated by the Fear of Recurrence Questionnaire (short form) - filled out by patients during follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Christian von Buchwald, Professor, MD, DMSci, Study Chair — Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Rigshospitalet
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery and Audiology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No